CLINICAL TRIAL: NCT01313364
Title: A Safety Study in Healthy Volunteers of the Single-Use Autoinjector Containing Placebo of BG9418 Interferon Beta-1a With a 25-Gauge × 1-Inch Needle
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The objective of the study has been achieved with fewer subjects than planned.
Sponsor: Biogen (Industry)
Responsible Party: Medical Director, Biogen Idec
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 108HV104
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects to self-administer 4 IM injections (Experimental): Subjects will be recruited and stratified into BMI groups: <18.5 kg/m2, 18.5 to 24.9 kg/m2, 25 to 29.99 kg/m2, and >30 kg/m2 all with 20 subjects. To maintain a balance between sexes that is representative of the MS population, approximately 50 to 70% of subjects within each BMI group should be female.
  Interventions: Device: 25G x 1" Needle Autoinjector

INTERVENTIONS:
Device: 25G x 1" Needle Autoinjector — All subjects will self-administer 4 IM injections using single-use autoinjectors.

SUMMARY:
This is a single-arm, single-center study in healthy volunteers. This study is designed to evaluate the safety of IM injections using single-use autoinjectors with a 25G × 1" needle. The purpose of this study is not to evaluate study treatment; therefore, all injections will be performed with Avonex placebo only; no active IFNβ-1a will be administered.

DETAILED DESCRIPTION:
This is a single-arm, single-center study in healthy volunteers. The study is designed to evaluate the safe use of the single-use autoinjector with a 25G × 1" needle in subjects of varying body mass indices (BMIs). Because this is a safety study of the injector, the injections contain Avonex excipients only; no active IFNβ-1a will be administered.

During the study, each subject will self-administer 4 IM injections using single-use autoinjectors.

Subjects will self-administer the first 2 injections (1 in each thigh) and then repeat the process approximately 60 to 90 minutes later. A Trainer/Observer will prepare the autoinjector for each injection, monitor each injection, and assess the subject for AEs during the injection process and up to the time of discharge from the unit. The Trainer/Observer will also visually inspect the needle pre- and post-injection and record their findings. The Investigator or designee (physician or nurse) will assess injection sites for erythema, induration, tenderness, or warmth.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females, aged 18 to 65 years, inclusive, at time of informed consent
* Able to understand and comply with the protocol
* Must be English or French speaking
* At the investigator's opinion, must be willing and able to perform self-injections into the right and left thighs with the single-use autoinjector

Exclusion Criteria:

* Abnormal screening blood tests determined to be clinically significant by the Investigator
* Treatment with any systemic anticoagulant within the previous 30 days
* Treatment with aspirin within the previous 7 days or nonsteroidal anti-inflammatory drugs (NSAIDs) within the previous 3 days
* History of severe allergic or anaphylactic reactions
* History of any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, pyschiatric, renal, and/or other major disease including bleeding disorders
* Current enrollment in any other investigational study
* Female subjects who are currently pregnant
* History of alcohol or substance abuse or a positive drug screening test on day 1

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent AEs reported when using the single-use autoinjector with a 25G x 1" needle | 24 hours

SECONDARY OUTCOMES:
Incidence (post-injection) of clinician-assessed injection site erythema, induration, tenderness, or warmth | 24 hours
Incidence of abnormal post-injection needle observations | 24 hours
Incidence of AEs associated with abnormal post-injection needle observations | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Toronto, Ontario, Canada